CLINICAL TRIAL: NCT04594070
Title: A Randomized Trial of Intermittent Oral Iron Supplementation vs. Daily Oral Iron Supplementation for the Treatment of Anemia in Pregnancy
Brief Title: Daily Versus Alternate Day Iron Supplementation for the Treatment of Iron Deficiency Anemia in Pregnancy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit enough participants
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-0068
Record Dates: First submitted 2020-09-30; First posted 2020-10-20 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Pregnancy Related; Iron Deficiency Anemia of Pregnancy
Keywords: Pregnancy; Iron deficiency; Anemia; Iron supplementation
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daily iron supplementation (Active Comparator): Oral ferrous sulfate, 325 mg, take once daily
  Interventions: Drug: Ferrous sulfate
- Alternate day iron supplementation (Experimental): Oral ferrous sulfated, 650mg, taken once daily every other day
  Interventions: Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Ferrous sulfate — Iron supplementation

SUMMARY:
The target population for our study is pregnant women in the first or second trimester with a diagnosis of iron deficiency anemia. If a subject is eligible, written consent will be obtained by person to person contact. Eligible participants will be randomized to receive either daily oral iron supplementation or every other day oral iron supplementation.

DETAILED DESCRIPTION:
Eligible pregnant women in the first or second trimester who carry a diagnosis of iron deficiency anemia as defined by the American College of Obstetrics and Gynecology will be approached, consented, and randomized to receive either daily oral ferrous sulfate (325mg) supplementation or every other day oral ferrous sulfate (650mg). Participants will undergo a phone survey 2-4 weeks after starting the study to assess for side effects. Participants will continue routine care and surveillance of iron deficiency in pregnancy until the end of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin less than 11 g/dl in the first trimester or less than 10.5 g/dl in the second trimester
* Microcytic anemia
* Singleton gestation in the first or second trimester

Exclusion Criteria:

* Malabsorptive disorder or history of restrictive or malabsorptive gastric surgery
* Known diagnosis of anemia other than iron deficiency (thalassemia, macrocytic, sickle cell, etc.)
* History of cardiopulmonary disease
* Severe anemia requiring parental infusion or transfusion of blood products

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 14 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melody Safarzadeh, MD, MS, Principal Investigator — UTMB
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol was terminated early due to low accrual.
Period: Overall Study
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Started | 8 | 6
Completed | 0 | 0
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Difference in Hemoglobin Levels From Enrollment to End of Study
Description: Hemoglobin levels will be assessed by blood draw upon enrollment and again in the third trimester of pregnancy
Time Frame: Baseline and again 8-9 months later (third trimester of pregnancy)
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Hematocrit in the Third Trimester After Treatment
Description: Hematocrit levels will be assessed by blood draw upon enrollment and again in the third trimester of pregnancy
Time Frame: Baseline and again 8-9 months later (third trimester of pregnancy)
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Gastrointestinal Side Effects After 2-4 Weeks of Treatment
Description: Gastrointestinal side effects with treatment will be assessed by telephone survey using a validated questionnaire.
Time Frame: 2-4 weeks after enrollment
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Complete Blood Count in the Third Trimester
Description: Complete blood count indices will be assessed by blood draw upon enrollment and approximately monthly until delivery
Time Frame: 8-9 months after enrollment (third trimester of pregnancy)
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Serum Ferritin at Time of Enrollment
Description: Serum ferritin will assessed by blood draw at time of enrollment.
Time Frame: Baseline only at time of enrollment
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Total Iron Binding Capacity at Time of Enrollment
Description: Total iron binding capacity will assessed by blood draw at time of enrollment.
Time Frame: Baseline only at time of enrollment
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Transferrin at Time of Enrollment
Description: Transferrin levels will assessed by blood draw at time of enrollment.
Time Frame: Baseline only at time of enrollment
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Receive Intravenous (IV) Iron Supplementation
Description: By chart review, we will determine if the subject received parental (IV) iron supplementation as part of the treatment for iron deficiency anemia
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Receive a Blood Transfusion
Description: By chart review, we will determine if the subject received a blood transfusion as part of the treatment for iron deficiency anemia
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Postpartum Hemoglobin
Description: Hemoglobin levels after delivery will be recorded (if obtained as part of regular postpartum care)
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Postpartum Hematocrit
Description: Hematocrit levels after delivery will be recorded (if obtained as part of regular postpartum care)
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Neonatal Weight at Delivery
Description: The weight of the baby (in grams) will be determined by chart review at the end of enrollment
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Level of Neonatal Bilirubin at Birth
Description: Neonatal hyperbilirubinemia will be reviewed and recorded by chart review
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Neonatal Apgar Scores
Description: Neonatal Apgar scores will be reviewed and recorded by chart review. The Apgar score is a method used to describe a newborn's status at birth and response to resuscitation. The Apgar score comprises five components: 1) color, 2) heart rate, 3) reflexes, 4) muscle tone, and 5) respiration, each of which is given a score of 0, 1, or 2. The range of scores is 0 to 10. Higher scores indicate reassuring newborn status.
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Newborns Who Are Admitted to the Neonatal Intensive Care Unit (NICU).
Description: The need for Neonatal Intensive Care Unit (NICU) Admission, will be assessed
Time Frame: At completion of study, on average after 9 months
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Weight Class at Time of Enrollment
Description: At time of enrollment the weight of the subject will be assessed and assigned a weight class using the World Health Organization weight classification
Time Frame: Baseline only at time of enrollment
Population: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No data collected due to early termination.
Description: No data collected due to early termination.
Arm/Group | Daily Iron Supplementation | Alternate Day Iron Supplementation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT04594070/Prot_SAP_000.pdf